CLINICAL TRIAL: NCT01808131
Title: A Long-Term Extension Study of Lesinurad in Combination With Allopurinol for Subjects Completing an Efficacy and Safety Study of Lesinurad and Allopurinol
Brief Title: Lesinurad and Allopurinol Combination Extension Study in Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDEA594-306; 2012-004389-16 (EudraCT Number)
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Gout
Keywords: Gout
MeSH Terms: conditions — Gout | interventions — lesinurad

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lesinurad 200 mg + allopurinol (Experimental)
  Interventions: Drug: Lesinurad
- lesinurad 400 mg + allopurinol (Experimental): Patients on lesinurad 400 mg had their dose changed to lesinurad 200 mg after implementation of protocol amendment 4, dated 07 October 2015.
  Interventions: Drug: Lesinurad

INTERVENTIONS:
Drug: Lesinurad — Tablets, 200 mg QD
  Arms: lesinurad 200 mg + allopurinol
Drug: Lesinurad — Tablets, 400 mg QD
  Arms: lesinurad 400 mg + allopurinol

SUMMARY:
This study will assess the serum uric acid lowering effects and safety of lesinurad in combination with allopurinol over a long-term timeframe.

DETAILED DESCRIPTION:
This is a Phase 3 extension study to assess the long-term efficacy and safety of lesinurad in combination with allopurinol in subjects who completed the double-blind treatment period in Studies RDEA594-301 and RDEA594-302.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the study procedures and the risks involved and is willing to provide written informed consent before the first study related activity.
* Subject completed the double-blind treatment period in either Study RDEA594-301 or RDEA594-302 and was actively receiving and tolerating study medication (lesinurad or placebo) and allopurinol at the Month 12 visit.
* Subject is male or female; female subjects of childbearing potential must agree to use an effective non-hormonal method of birth

Exclusion Criteria:

* Subject has any medical or psychological condition, which in the opinion of the Investigator and/or the Medical Monitor, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements, or to complete the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 717 (Actual)
Dates: Start 2013-02; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an sUA level that is < 6.0 mg/dL | up to a total of 5 years

SECONDARY OUTCOMES:
Resolution of at least 1 target tophi | Up to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Nihar Bhakta, MD, Study Director — Ardea Biosciences, Inc.
Locations (182):
- United States (128):
  - Birmingham, Alabama
  - Gulf Shores, Alabama
  - Pinson, Alabama
  - Glendale, Arizona
  - Mesa, Arizona
  - Peoria, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Gold River, California
  - Irvine, California
  - Roseville, California
  - Sacramento, California
  - San Diego, California
  - San Leandro, California
  - San Ramon, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Englewood, Colorado
  - Brandon, Florida
  - Brooksville, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Miami, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Plant City, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Conyers, Georgia
  - Johns Creek, Georgia
  - Roswell, Georgia
  - Savannah, Georgia
  - Honolulu, Hawaii
  - Idaho Falls, Idaho
  - Meridian, Idaho
  - Gurnee, Illinois
  - Cedar Rapids, Iowa
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Paducah, Kentucky
  - Metairie, Louisiana
  - Natchitoches, Louisiana
  - Cumberland, Maryland
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Flint, Michigan
  - Kalamazoo, Michigan
  - Southfield, Michigan
  - Traverse City, Michigan
  - Hazelwood, Missouri
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Washington, Missouri
  - Omaha, Nebraska
  - Reno, Nevada
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Hartsdale, New York
  - New York, New York
  - Calabash, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Shelby, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Colombus, Ohio
  - Dayton, Ohio
  - Franklin, Ohio
  - Middleburg Heights, Ohio
  - Perrysburg, Ohio
  - Willoughby Hills, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Altoona, Pennsylvania
  - Clairton, Pennsylvania
  - Duncansville, Pennsylvania
  - Indiana, Pennsylvania
  - Jenkintown, Pennsylvania
  - McMurray, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Scottdale, Pennsylvania
  - Columbia, South Carolina
  - Mt. Pleasant, South Carolina
  - Myrtle Beach, South Carolina
  - Rock Hill, South Carolina
  - Spartanburg, South Carolina
  - Union, South Carolina
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Spring Hill, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Irving, Texas
  - Kingwood, Texas
  - Nassau Bay, Texas
  - Plano, Texas
  - San Angelo, Texas
  - San Antonio, Texas
  - Sealy, Texas
  - Sugar Land, Texas
  - Waco, Texas
  - Bountiful, Utah
  - Layton, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Danville, Virginia
  - Manassas, Virginia
  - Midlothian, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Olympia, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Australia (5):
  - Herston, Queensland
  - Clayton, Victoria
  - Heidelberg West, Victoria
  - Brisbane
  - Woodville South
- Belgium (4):
  - Genk
  - Kortrijk
  - Lommel
  - Yvoir
- Canada (6):
  - Coquitlam, British Columbia
  - Penticton, British Columbia
  - Kitchener, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Québec, Quebec
- Germany (5):
  - Eichstätt, Bavaria
  - Goch, North Rhine-Westphalia
  - Dresden, Saxony
  - Kamenz, Saxony
  - Leipzig, Saxony
- New Zealand (7):
  - Grafton, Auckland
  - Otahuhu, Auckland
  - Beckenham, Christchurch
  - Birkinhead
  - Hamilton
  - Rotorua
  - Tauranga
- Poland (6):
  - Poznan, Greater Poland Voivodeship
  - Krakow, Lesser Poland Voivodeship
  - Katowice, Silesian Voivodeship
  - Warminsko-mazurskie
  - Warsaw
  - Gmina Końskie, Świętokrzyskie Voivodeship
- South Africa (14):
  - Newlands, Durban
  - Silverglen, Durban
  - Newtown, Johannesburg
  - Parktown, Johannesburg
  - Radiokop, Johannesburg
  - Sowento, Johannesburg
  - Thabazimbi, Limpopo
  - Muckleneuk, Pretoria
  - Durban
  - Paarl
  - Rondebosch
  - Stellenbosch
  - Witbank
  - Worcester
- Spain (2):
  - Mérida, Badajoz
  - A Coruña
- Lausanne, Canton of Vaud, Switzerland
- Ukraine (4):
  - Kharkiv
  - Kyiv
  - Poltava
  - Vinnytsia